CLINICAL TRIAL: NCT06488872
Title: Comparison of Artificial Intelligence-based Analysis of Computed Tomography Data With Routinely Performed Measurements Concerning Bone and Muscle Health of Aged Individuals to Validate Surrogate Parameters for the Aging Population.
Brief Title: Comparison of Computed Tomography Data With Routine Measurements Concerning Bone and Muscle Health of Aged Individuals
Acronym: SARCATAR
Status: Recruiting | Type: Observational
Sponsor: University Department of Geriatric Medicine FELIX PLATTER (Other)
Responsible Party: Principal Investigator, Andreas Fischer, PD Dr.med. Andreas M. Fischer, Principal Investigator, Head of NutriCare Clinic, University Department of Geriatric Medicine FELIX PLATTER
Other Study IDs: 2024-0705
Record Dates: First submitted 2024-06-18; First posted 2024-07-05 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Sarcopenia; Muscle Loss; Osteoporosis
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: comparison of CT scan with routinely assessed methods of muscle mass and strength — comparison of CT scan with routinely assessed methods of muscle mass and strength

SUMMARY:
This study focuses on researching sarcopenia and bone loss (osteoporosis), aiming to develop early and effective methods for diagnosis and treatment. These health issues significantly contribute to falls, fractures, and loss of independence and quality of life in old age, particularly affecting individuals impairments. To address these challenges, the study employs innovative imaging techniques based on artificial intelligence (AI) to accurately assess age-related muscle atrophy. A central approach is to analyze existing computed tomography (CT) images of older adults, using retrospective data to evaluate muscle quality. This method aims to efficiently assess muscle quality without additional resources. AI algorithms analyze fine details of muscle tissue, such as muscle adiposity and density. The algorithm can detect fat content within muscles, which negatively impacts muscle health and functionality, and identify irregularities or abnormalities in muscle fibers. This non-invasive approach is crucial for early detection of muscle atrophy and monitoring treatment success. Integrating AI technologies advances beyond conventional imaging techniques, allowing precise analysis of muscle quality. This method not only offers efficient diagnosis and monitoring of sarcopenia but also opens new avenues for personalized therapeutic approaches and improved patient care. Almost every elderly person has at least one existing CT scan, a common and excellent method of medical imaging for significant health issues. These images can be retrospectively analyzed for muscle health. In addition to imaging techniques, the study includes functional tests such as hand strength and walking speed measurements to assess muscle health and condition. These tests establish objective quality characteristics of muscles and assess the effectiveness of prevention and treatment measures. This research aims to provide early diagnosis and effective treatment strategies for sarcopenia and osteoporosis, ultimately improving the quality of life for the elderly. By leveraging AI and existing medical imaging data, the study promotes efficient, sustainable, and precise healthcare solutions for age-related muscle and bone deterioration.

DETAILED DESCRIPTION:
Age-related muscle wasting and bone loss are significant public health challenges impacting elderly mobility and independence. Sarcopenia, a decline in muscle strength and mass, heightens fall risk, particularly in individuals with dementia or cognitive impairments. This leads to complications, reduced independence, and diminished quality of life. Osteoporosis increases the risk of fractures from falls or spontaneously, necessitating early diagnosis and prevention.

Despite effective treatments for sarcopenia, such as a protein-rich diet and strength training, the condition remains underrecognized due to diagnostic challenges. Common methods like hand strength measurement are problematic for those with rheumatic conditions or Parkinson's, often yielding inaccurate results. Other methods, like measuring leg strength and walking speed, require coordination and balance, which can be difficult for those with dementia or visual impairments. There is a need for tailored diagnostic solutions for diverse aging populations.

Bone mineral density (BMD) is crucial for assessing health in older adults, as low BMD indicates osteoporosis and a higher fracture risk. Traditionally measured by dual X-ray absorptiometry (DEXA), BMD assessment can be difficult for patients with mobility issues, pressure ulcers, or dementia due to the requirement to remain still for extended periods.

New AI-based algorithms can now automatically evaluate body tissues and patterns from routine CT scans, offering reproducible results beyond human capability. AI can quantify muscle mass at specific body cross-sections, such as lumbar vertebral point 3 (L3), which correlates with total body muscle mass and predicts muscle health. CT measurements of thigh and psoas muscles can also indicate whole body skeletal muscle mass. European guidelines highlight the need for muscle quantification in early sarcopenia diagnosis.

Correlating AI-measured muscle mass with functional muscle strength assessments can help identify surrogate parameters for early sarcopenia detection. Additionally, measuring muscle fat content, which correlates with strength loss, is essential for assessing muscle health. Innovative approaches are required, as sarcopenia diagnosis is still evolving and geriatric diseases often need proportionate diagnostic and treatment strategies due to multiple comorbidities.

For osteoporosis diagnostics, AI can determine Hounsfield Unit (HU) values from CT images to represent bone density, which can be correlated with DEXA results. These surrogate diagnostics should follow current guidelines, with results obtained within an appropriate interval of up to 18 months.

Based on the primary endpoints, the prevalence of "muscle-healthy" and "probably sarcopenic" individuals will be recorded. Additionally, the prevalence of individuals without osteoporosis, with osteopenia, and with confirmed osteoporosis will be calculated and included in the analysis.

The secondary endpoints compare functional muscle strength measurements with retrospective quantitative CT results. This exploratory analysis will test whether the AI algorithm can correlate functionality with muscle volume. Additionally, AI-measured muscle fatness (myosteatosis) could serve as a new, quantifiable quality criterion for muscle health. This is important because many elderly individuals cannot meet functional strength test requirements due to conditions like visual impairment, dementia, chronic pain, joint diseases, and frailty.

For osteoporosis diagnostics, the investigators aim to correlate bone density from DEXA measurements with CT-derived bone density of thoracic and abdominal vertebral bodies. This exploratory surrogate measurement method could provide insights into bone mineral density and health from existing CT images. CT-based diagnosis could be an alternative for those unable to remain still for DEXA scans.

Design:

This retrospective study will be conducted at a single center. Participants will be identified using databases of patients who have undergone CT and DEXA scans. To be included in the sarcopenia arm, participants must have had a CT scan from the radiology department at the University Hospital Basel within one month of an inpatient stay. For the osteoporosis arm, a thorax and/or abdomen CT scan and a DEXA scan must be available, conducted within 18 months of each other.

Anonymized DICOM datasets from the CT scans will be analyzed by an AI algorithm. Data analysis will involve standard statistical comparison using Student's t-test. The algorithm's values will be tested against reference standards, and its diagnostic accuracy will be evaluated for various diseases. The algorithm has been tested on 104 anatomical structures, organs, and organ groups (Req-2022-00495).

Origin of the data:

At the largest geriatric medical center in Switzerland, the investigators would like to include geriatric patients aged 65 and over who were undergoing inpatient treatment in the period from 01.07.2017 to 31.12.2022 inclusive.

By testing alternative diagnostic procedures (exploratory approach), the investigators want to reach more people, especially those who are unable to follow current diagnostic procedures due to dementia, visual impairment or post-operative condition. This is crucial as these patients in particular have a significantly increased risk of falling. The research approach aims to address real-world challenges in order to consider prevention programs and personalized therapies for as many people as possible in the future.

By using existing data and dispensing with further investigations, the economic aspect in the context of rising healthcare costs is also taken into account.

Scientific methodology and targets:

Exploratory analysis of quantitative variables that can be determined by CT to evaluate the primary endpoints:

* Sarcopenia: By evaluating muscle volume and fat percentage in muscle (in mm3) and density (in HU) on CT.
* Osteoporosis: By evaluating bone density/attenuation in HU on CT. For the evaluation of muscle volumes and densities, a feasibility study has already been carried out on a representative sample of over 4000 patients, which suggests a normal distribution of muscle density and volume (21). Statistical deviations from this reference group are determined using a t-test or Wilcoxon test in the case of a lack of normal distribution. The test for normal distribution is performed using the Kolmogorov-Smirnov test. The significance level is set at α = 0.05.

The evaluation of osteoporosis is performed analogously. The relationship between attenuation in HU and BMD has already been documented in the literature (22) (18).

Inclusion of as many patients as possible is essential for representative results

For which health-related personal data should consent be granted? A general consent form "Declaration of consent for the further use of health-related data and samples" was introduced at the beginning of 2020. Unfortunately, in practice it proved to be unreasonable to implement.

The investigators consider the sample size to be n=300. No consent has been obtained for any of the participants, meaning that an application for exemption is being made for all persons.

Quantitative, clinical data:

Hand strength measurement on both hands (geriatric routine assessment to assess the muscle strength of the upper extremity)

* Gait speed (geriatric routine assessment to assess mobility and muscle strength of the lower extremity; important for predicting falls)
* Timed up & go (geriatric routine assessment to assess muscle strength of the lower extremity, coordination and sense of balance; important for predicting falls)
* Vitamin D level in serum (underestimated vitamin in old age, which is produced by the body itself through natural sunlight exposure of the skin and good kidney function in the investigators latitudes through many intermediate steps and contributes significantly to bone and muscle health; in the investigators latitudes (angle of incidence of the sun's rays), sufficient vitamin D production is only possible in the months of April to October with sufficient time spent outdoors. With age, however, the ability to synthesize vitamin D production also decreases considerably in the spring to summer months.

Quantitative data from imaging:

* Previous DEXA measurements of bone density (T-score, Z-score)
* Muscle mass and fat content in the muscle from previous CT scans (thorax, abdomen, pelvis, spine with muscle parts shown)

ELIGIBILITY:
Inclusion Criteria:

* CT examination (thorax, abdomen, pelvis, spine with muscle parts to be visualized) by the responsible in-house radiology department one month before or after the inpatient stay at the UAFP (sarcopenia arm).
* CT thorax and CT abdomen images of patients from the responsible in-house radiology department and an in-house DEXA measurement. Both examinations may be performed no more than 18 months apart (osteoporosis arm).
* Diagnostic image quality of CT scans.

Exclusion Criteria:

* Presence of a documented refusal.
* Non-diagnostic image quality
* Absence of the following functional measurements: Hand strength on both hands, timed-up & go test, gait speed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We would like to retrospectively examine a total of 300 data sets of geriatric patients from 01.01.2017 to 31.12.2022, who were treated as inpatients at the UAFP. Individuals will be identified using various databases containing information on patients who have undergone CT scans imaging the thoracic and/or abdominal organs and DEXA scans.
  Participants must have had a CT scan performed by the in-house radiology department one month before or after the inpatient stay.
  In order to be included in the osteoporosis arm, a thorax and/or abdomen CT scan and a DEXA scan from an in-house DEXA measurement must be available. Both examinations must not be more than 18 months apart.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Volume in mm3 on CT | through study completion, an average o 1 year
  Exploratory analysis of quantitative variables that can be determined by CT to evaluate the primary endpoint Sarcopenia: By evaluating muscle volume (in mm3) on CT.
fat percentage in muscle density (in HU) on CT. | through study completion, an average o 1 year
  Exploratory analysis of quantitative variables that can be determined by CT to evaluate the primary endpoint Sarcopenia: By evaluating fat percentage in muscle density (in HU) on CT.
bone density/attenuation in HU on CT. | through study completion, an average o 1 year
  Analysis of bone density/attenuation in HU on CT to evaluate the primary endpoint Osteoporosis:

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M. Fischer, PD Dr., Principal Investigator — Universitäre Altersmedizin Felix Platter
Locations (1):
- Universitäre Altersmedizin Felix Platter, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372